CLINICAL TRIAL: NCT03565796
Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2018: a Single-blind Cluster Randomized Controlled Trial on Brief Intervention (AWARD), Active Referral and Financial Incentive for Attending Smoking Cessation (SC) Service to Increase Abstinence
Brief Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QTW 2018
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Quit to Win; Brief intervention; Financial incentive; Active referral; AWARD model
MeSH Terms: conditions — Smoking Cessation | interventions — corticosteroid hormone-induced factor; Referral and Consultation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Personalized active referral plus financial incentive+ AWARD advice + referral card + warning leaflet+ COSH booklet
  Interventions: Behavioral: Personalized active referral plus financial incentive; Behavioral: AWARD advice; Behavioral: Warning leaflet; Behavioral: Referral card; Behavioral: COSH booklet
- Group B (Experimental): AWARD advice + COSH booklet
  Interventions: Behavioral: AWARD advice; Behavioral: COSH booklet

INTERVENTIONS:
Behavioral: Personalized active referral plus financial incentive — Smokers will be introduced to various SC services in Hong Kong and be motivated to use the services.Written consents will be obtained from smokers who are ready to book the service onsite for transfer of their contact telephone numbers to their chosen service providers. Our research staff will transfer the information to the service providers within a week since the enrollment.Smokers are informed at baseline that they will receive financial incentive (supermarket coupon HK$300) if they attend or use any of the SC services within 3-month.
  Arms: Group A
Behavioral: AWARD advice — Ask about smoking history, Warn about the high risk of smoking, Advise to quit as soon as possible, Refer to the smoking cessation services, and Do it again (if the smokers refused to set quit date).
  Other Names: Ask, Warn, Advise, Refer, Do-it-again
Behavioral: Warning leaflet — The 2-sided color printed A4 leaflet, which systematically covers the most important messages to motivate smoking cessation
  Other Names: Brief leaflet on health warning and smoking cessation
  Arms: Group A
Behavioral: Referral card — The 3-folded "Smoking Cessation Services" card consists of brief information and highlights of existing smoking cessation services, contact methods, motivation information and strong supporting messages or slogans
  Other Names: Smoking Cessation Service Card
  Arms: Group A
Behavioral: COSH booklet — A general smoking cessation self-help booklet
  Other Names: COSH self-help smoking cessation booklet

SUMMARY:
The present study will examine (1) the effectiveness of a combined intervention of face-to-face brief cessation advice (AWARD), active referral of SC service plus financial incentive on encouraging SC services use and (2) explore the use of CBPR model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, a process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

DETAILED DESCRIPTION:
Although smoking prevalence is decreasing in Hong Kong, there are still 615,000 daily cigarette smokers in Hong Kong in 2017 and half will be killed by smoking which accounts for over 7,000 deaths per year. Smoking also accounts for a large amount of medical cost, long-term care and productivity loss of US$688 million (0.6% Hong Kong GDP). Smoking is a highly addictive behavior and it is difficult for smokers with strong nicotine dependence to quit without assistance. On the other hand, reaching and helping the many smokers who have no intention to quit is a challenge, because they are unlikely to seek professional help from smoking cessation services.

The Quit and Win programme provides an opportunity to reach and encourage a large group of smokers to make quit attempt and maintain abstinence. The Quit and Win model posits that smokers participating in the contest will have higher motivation to quit with incentives and better social support. Studies have found that such quitting contests or incentive programs appeared to reach a large number of smokers and demonstrated a significantly higher quit rate for the quit and win group than for the control group.

SC services utilization rates are markedly low in Hong Kong. The latest Thematic Household Survey reported that only 3.3% daily smokers had ever used SC services. Among never-used smokers, only 3.1% of them were willing to try the SC services. The previous trial in QTW Contest 2016 depicts a similar pattern. Despite over three quarters of participants (77.0%) in the HAR group had chosen an SC service. Among them, only a small percentage (34.9%) actually used the SC service. Most smokers (65.1%) failed to attend the SC service under the HAR intervention. Consequently, better interventions are needed to extend the reach of SC services and smokers who had chosen an SC service but fail to attend.

The previous trial in QTW Contest 2013 showed a small cash incentive with early notifications increased quit attempt by self-directed help, but it did not increase abstinence and the use of formal cessation aids. Therefore, financial incentive-based SC programme focusing on promoting existing SC services use is warranted.

Therefore, the present study will examine (1) the effectiveness of a combined intervention of face-to-face brief cessation advice (AWARD), active referral of SC service plus financial incentive on encouraging SC services use and (2) explore the use of CBPR model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, a process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 cigarette per day in the past 3 months
* Able to communicate in Cantonese (including reading Chinese)
* Exhaled carbon monoxide (CO) 4 ppm or above, assessed by a validated CO smokerlyzer
* Intent to quit / reduce smoking

Exclusion Criteria:

* Smokers who have difficulties (either physical or cognitive condition) to communicate
* Currently following other smoking cessation programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1093 (Actual)
Dates: Start 2018-06-16 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Biochemical validated quit rate | 3-month follow-up
  The primary outcomes are biochemically validated quit rates at 3-month in the two groups
Biochemical validated quit rate | 6-month follow-up
  The primary outcomes are biochemically validated quit rates at 6-month in the two groups

SECONDARY OUTCOMES:
Smoking quit rate change from baseline at 3-month follow-up | 3-month follow-up
  Self-reported 7-day point prevalence (pp) quit rate at 3-month between the two groups
Smoking quit rate change from baseline at 6-month follow-up | 6-month follow-up
  Self-reported 7-day point prevalence (pp) quit rate at 6-month between the two groups
Smoking reduction rate change from baseline at 3-month follow-up | 3-month follow-up
  Rate of smoking reduction by at least half of baseline amount in the two groups
Smoking reduction rate change from baseline at 6-month follow-up | 6-month follow-up
  Rate of smoking reduction by at least half of baseline amount in the two groups
Smoking quit attempt change from baseline at 3-month follow-up | 3-month follow-up
  Number of quit attempts at 3-month in the two groups
Smoking quit attempt change from baseline at 6-month follow-up | 6-month follow-up
  Number of quit attempts at 6-month in the two groups
Quit rate for all subjects change from baseline at 3- and 6-month follow-up | 3 and 6 months follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2018
Reduction rate for all subjects change from baseline at 3- and 6-month follow-up | 3 and 6 months follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2018
Use of smoking cessation service | 3 and 6 months follow-up
  Use of smoking cessation at 3 and 6 month follow-up in the two groups
Use of smoking cessation service for all subjects | 3 and 6 months follow-up
  Use of smoking cessation service for all subjects participating in Quit to Win contest 2018

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Kelvin Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong Council on Smoking and Health (COSH), Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weng X, Wu Y, Luk TT, Li WHC, Cheung DYT, Tong HSC, Lai V, Lam TH, Wang MP. Active referral plus a small financial incentive upon cessation services use on smoking abstinence: a community-based, cluster-randomised controlled trial. Lancet Reg Health West Pac. 2021 Jul 5;13:100189. doi: 10.1016/j.lanwpc.2021.100189. eCollection 2021 Aug. PMID 34527982
- [Derived] Weng X, Wang MP, Li HCW, Cheung YTD, Lau CY, Kwong ACS, Lai VWY, Chan SSC, Lam TH. Effects of active referral combined with a small financial incentive on smoking cessation: study protocol for a cluster randomised controlled trial. BMJ Open. 2020 Oct 26;10(10):e038351. doi: 10.1136/bmjopen-2020-038351. PMID 33109654
- [Derived] Luk TT, Weng X, Wu YS, Chan HL, Lau CY, Kwong AC, Lai VW, Lam TH, Wang MP. Association of heated tobacco product use with smoking cessation in Chinese cigarette smokers in Hong Kong: a prospective study. Tob Control. 2021 Nov;30(6):653-659. doi: 10.1136/tobaccocontrol-2020-055857. Epub 2020 Sep 10. PMID 32912861